CLINICAL TRIAL: NCT03641001
Title: Impact of Nutrition Intervention (Counselling, Food Voucher for Recipe, WASH and Home Fortification) on Growth and Feeding Practices of Under Two Years Children in Rural Bangladesh"
Brief Title: Nutrition Intervention Integrated With Food Voucher to Improve Child Growth and Feeding Practices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Brac (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-17083
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Child Malnutrition; Feeding Behavior; Growth; Stunting, Nutritional
Keywords: Intervention; Food voucher; Child feeding; Growth; WASH
MeSH Terms: conditions — Child Nutrition Disorders; Feeding Behavior; Growth Disorders | interventions — Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: Community based Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group will receive child feeding counselling, food voucher for recipe, WASH and home fortification
  Interventions: Behavioral: Child feeding counselling, food voucher, micronutrient powder, WASH
- Control (No Intervention): Control will receive usual health messages from government and NGO

INTERVENTIONS:
Behavioral: Child feeding counselling, food voucher, micronutrient powder, WASH — Child feeding counselling will be assisted by food voucher, micronutrient powder and WASH messages
  Arms: Intervention

SUMMARY:
Brief Summary: Background:

The period from birth to two years of age is the "critical window" for the promotion of optimal growth, health, and development. Insufficient quantities and inadequate quality of complementary foods, poor child-feeding practices and high rates of infections have a detrimental impact on growth. Approximately one-third of children less than 5 years of age in developing countries are stunted, and large proportions are also deficient in one or more micronutrients. An estimated 6% or 6 hundred thousand under-5 deaths can be prevented by ensuring optimal complementary feeding (CF) only.

Knowledge gap:

Even though the importance of CF is established, children < 2y are being fed complementary foods with poor nutrient quality, particularly in resource poor countries like Bangladesh.

Relevance:

Approximately 36% under 5 children are stunted in Bangladesh. Only 23% of children age 6-23 months is fed appropriately based on recommended infant and young child feeding (IYCF) practices. The routine diet of the population including children is mainly plant based and lacks adequate protein and other essential nutrients. Hygiene is also an issue as only 21% of rural households use soap and water during handwashing. An intervention package including CF counselling, WASH and micronutrient powder (MNP) could be potential option for optimizing complementary feeding practice in rural Bangladesh.

Hypothesis: An integrated intervention package will improve child growth in terms of length and complementary feeding practice in the selected intervention area from rural Bangladesh compared to control area.

Objectives:

1. To improve nutritional status (length for age Z-score or LAZ) of the children (6-12 mo) through food voucher to promote improved recipe and intervention package with 12 months of intervention period.
2. To improve young child feeding practices following counselling

Methods:

This will be a community based cluster randomized trial. Group I (intervention) will receive a package of intervention (child feeding counselling, WASH and micronutrient powder) along with food voucher to support feeding their children a homemade snack following a newly developed recipe (suzi firni for <1 year, suzi halua for >1 yr) and Group II (Control) will receive usual health meassages. Baseline and endline survey will be conducted. Growth Monitoring Promotion (GMP) will be done monthly to monitor the growth of the children and utilization of food voucher. Data on child feeding, morbidity and anthropometry (length and weight) will be collected monthly.

Outcome measures/variables:

1. Difference in mean LAZ of the children between intervention and control group
2. Difference in mean weight for age Z-score (WAZ) of the children between intervention and control group
3. Difference in proportions of mothers in terms of correct knowledge and practice on CF

DETAILED DESCRIPTION:
Study design We will use a cluster randomized study design with cross-sectional surveys at baseline and endline to examine the effect of an integrated intervention package consisting of BCC, food voucher system to feed the children homemade snack following a recommended recipe, MNP and tailor-made counselling on hand washing and food safety to improve child growth and feeding practices. The effect of the intervention package will be compared to a control group which will be an adjacent area (see diagram) with similar population demography receiving usual health messages. The primary outcome assessment will be done through comparing differences in nutritional status of the children (<2y) among intervention and control groups. Also the change in knowledge, attitude and practice (KAP) regarding child feeding practices among mothers from intervention and control groups will be assessed.

Study site and participants The study will be conducted in Harirumpur sub-districts of Manikgonj. The study area is selected purposively in consultation with brac considering transportation and logistical issues. The Harirumpur sub-district has 13 unions and out of these, 3 unions will be selected randomly for intervention and the 3 unions will serve as control group (Control Group l). Random allocation of the intervention will be performed by a scientist from icddr,b who will not be involved with this study.

Inclusion criteria for study participants

1. Households having under two years children (6-12 mo during enrolment)
2. Household listed as poor household following above mentioned criteria
3. Not involved with any government/non-government microfinance programme
4. Not participants of any IYCF programme Components of the intervention package The intervention package includes-

1. BCC on child feeding practices 2. Food voucher to support feeding of a homemade snack (suzi Firni/Halua) and the recipe will be demonstrated to the mothers by SS and Pushti kormi (PK) in group sessions 3. Regular WASH messages PLUS new messages on risk and management of poultry faeces 4. Home-based fortification with MNP Description of the intervention package

Development of Behaviour Change Communication (BCC) materials:

Behaviour change communication (BCC) is an interactive process of any intervention with individuals, communities and/or societies (as integrated with an overall programme) to develop communication strategies to promote positive behaviours which are appropriate according to the context. This in turn provides a supportive environment that enables people to initiate, sustain and maintain positive and desirable behaviour. SSs and PK will use existing harmonized BCC tools (child feeding counselling packages including flip chart, videos) to inform mothers regarding optimum child feeding practice. However, considering the objectives of the proposed study some additional materials will be developed. The major topic of the BCC materials will be promotion of newly developed recipe and WASH. Adequate and clear message will be delivered to the mother regarding the new recipe so that it should be treated as snack only and must not replace any major meal of the day.

Food voucher conditional on practicing recommended recipe:

Each of the mothers of under two years children ( 6-12 mo) will receive voucher as coupon or piece of paper that can be exchanged for goods. The Vouchers will allow the mothers to purchase commodities for Suzi recipe from the participating vendors without using of cash. Participating vendors will be selected according to predetermined criteria. A mother will be given a voucher equivalent to a certain amount of cash which she can spend at any pre-approved vendor. A voucher will have to be spent out within a certain time period before becoming invalid ("redemption period") to maintain compliance which will be monitored by research staff. It is expected that this type of voucher will offer us to have control over the purchase of items and its use, because of the programmatic reason we need to restrict purchases to a specific, identified food commodity to feed the children.

brac will provide monthly food voucher equivalent to BDT, 1100 (proposed) to feed prescribed snack recipe to their children in order to ensure daily consumption of some animal source protein and added energy along with their regular diet. The sole purpose of the food voucher is to improve dietary diversity of the children in the intervention areas. The amount of food voucher is estimated on monthly basis considering associated cost of buying all the ingredients for cooking of "Suzi firni/ halua" which should be consumed two times per day as snacks. Some of them, however, may have internal arrangement of serving this proposed food from their own capacity; in such case they will be suggested/encouraged to spend this food voucher to exchange nutritious complementary food especially animal protein for their children.

Monthly feeding history, morbidity as well as anthropometric data of the children will be collected by the data collection tream of icddr,b. If it is reported that someone among the children from intervention group is not gaining weight in subsequent months, investigators will try to find out the valid reason. If required, the children will be referred to the local government, NGO or private hospital for further follow up for better diagnosis.

Home fortification:

The SS will distribute one-month supply of micronutrient powder (MNP) during home visits once at a time in the intervention group. A zip-lock bag will be provided to every mother to store the empty sachets to ensure compliance. Mothers will be asked to add MNP with complementary food. SS will demonstrate mothers to mix MNP with main meal by dividing the meal into two parts and mix the whole sachet of MNP with one portion and feed the MNP mixed part of food first and then the next portion. By using counselling card, they will provide instruction to feed MNP mixed food within half an hour to avoid metallic taste and also inform to use one sachet for one child. A child will be given at least 10 sachets at every month followed by 60 sachets in six months and 120 sachets in a year.

Child WASH:

Hygienic practices and hand washing will be one of the major areas to counsel mother in terms of hand washing before food preparation, before and after child feeding and defecation. Frontline workers (SS & PK) will advise the mothers and caregivers to maintain personal hygiene e.g. cutting nails, use of footwear, washing hand before preparing food and feeding their children for prevention of infection and worm infestations during their routine visits. The SS and PK will provide tailored messages on hand washing focusing on sanitation and clean environment specially protecting child from ingestion of poultry feces, safe disposal of child feces, safe drinking water (collection, transport, storage, treatment). To inform and educate mothers regarding the hazardous effect of ingestion of poultry faces and subsequent environmental enteropathy, materials will be developed namely "CHILD WASH". Till date no such BCC material is reported in the country; therefore existing BCC materials on WASH used by government, development partner, local and international NGOs and used in other countries will be reviewed by IYCF experts and BCC martial specialist. According to their comments and opinions, draft BCC materials will be designed by a contracted agency. The draft materials will be tested in the field to find out its comprehensibility, clearness of the content by the mothers and caregivers in community setting. Pilot testing will not include the households those are included in the original study. Necessary changes will be done on the basis of feedback from field testing. The SS and PK will receive training on these newly developed materials so that they can deliver the message clearly and concisely to encourage mothers to adopt the practice. The control group will receive regular WASH messages focusing on hand washing and use of safe water.

Home visits by SS and PK Scheduled home visits are carried out by SS and PK. SS registers all children 0-2 years in her area and visits at least once a month to counsel and demonstrate techniques of continuation of breastfeeding up to 24 months. During this study, special emphasis will be given on CF in terms of new recipes (Suzi firni/ halua), homemade complementary food, appropriate amount and frequency of complementary foods and consumption of protein from animal source according to age for children 7-24 months. Mothers will be advised to utilize the voucher to purchase ingredients for proposed recipe to feed her child by following any of the recipes according to her convenience. Importance will be given on hygiene and handwashing practice as well. Fortnightly courtyard session will be organized by SS and PK with a group of 10-12 mothers of study children for group counselling and practical demonstration of hand washing aid.

Acceptability of the new recipe:

The acceptability of the new recipe will be conducted among 50 children and their respective mothers/caregivers. The mothers will be requested not to give/allow any food and breast milk during the preceding 2 hours of observed meal time on the day of feeding observation which will be done under the direct supervision of trained study staff (2 observations). The feeding episode will last for maximum 60 minutes. The mothers will be asked to spoon feed their children the pre-weighed diet until the child refuses to eat further. Children will be considered as refusing further intake if they move their head away from the food, cry, clamp the mouth or clinch the teeth, or become agitated, spit out the food or refuse to swallow. The amount of food actually ingested will be calculated by subtracting the left over from the offered amount. Pre-weighed napkins will be provided; any food that is regurgitated, vomited or spilled will be swabbed, weighed and subtracted from the amount offered.

Acceptability will be categorized as 'accepted eagerly' if they ate food readily, did not make a fuss, spit out, vomit or cry during the observed meal. Children will be categorized as 'accepted but not eagerly' if they ate the offered food but either made fuss, spit out, vomited or cried during the observed meal. The third category will be children who will not consume the offered food at all. Perception and assessment of organoleptic characteristics (color, smell, taste, texture, etc.) of the prepared recipe by the respective mother/caregiver will also be assessed by using the 9-point Hedonic scale Intervention period: 12 months to ensure there is sufficient time to measure the IYCF practices and child growth.

Process evaluation:

To assess the fidelity of the program implementation, process evaluation will be carried out focusing on the program's operations, implementation, and service delivery. The process evaluation will identify the legibility of selecting study participants, implementation of voucher system, use of voucher, quality of the different awareness sessions carried out by SS and PK, satisfaction of the people involved in program implementation and probable challenges. Qualitative interviews, focus groups with the intervention recipients and family members (women, husbands, mothers-in-law), and implementers (i.e. project staff, SS/ PK/ PO, participating in the project) will be conducted.

Timeline for data collection: Information regarding process evaluation will be collected once in every 1 month.

Measurements Sample Size Calculation and Outcome (Primary and Secondary) Variable(s) To observe a difference of 0.4 in mean LAZ between intervention and control group (-1.4 vs -1.8, standard deviation 1.2) after 12 months intervention period, using a two-tailed t-test, a power of 80%, a significance level of 5%, and design effect of 1.3, the sample size for one arm is calculated = 184. With 10% attrition, the final sample size for intervention or control arm is 205 so the total sample size will be 205*2= 410 mother-child pairs.

Data Analysis Analyses will be conducted at the mother-infant dyad level, but will be adjusted for the community-cluster randomization. The primary analyses will compare the mean difference of LAZ in children after 12 months of intervention period using independent sample t- test and 95% confidence intervals for the group difference, adjusted for clustering. We will report the results for 2-sided 5% tests for the primary trial outcome. Secondary analyses will examine each outcome variable (minimum meal frequency, minimum dietary diversity, minimum acceptable diet, weight-for-age, maternal knowledge) taking account of the repeated measurements within children by using separate mixed models. We will use linear mixed models for continuous outcomes (e.g. length-for-age Z) and generalized linear mixed models for non-continuous outcomes (e.g. logistic mixed models for binary outcomes e.g. percentage with minimum dietary diversity). Models will include treatment group as a fixed effect, infants as a random effect to account for the repeated measurements, and community-cluster as a random effect to account for the cluster effect.

The models will be able to evaluate the impact of the interventions over time by testing for an interaction between time and intervention group. Analyses will be conducted to identify the baseline characteristics of mother-infant dyads who may benefit most from the intervention. Model assumptions will be checked and appropriate adjustments to the analysis will be made where necessary. STATA® software will be used for all analyses, with xtmixed command to fit linear mixed models and xtmelogit command to fit mixed-effects models for binary outcomes/responses. Also difference in differences analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Households having under two years children (6-12 mo during enrolment)
* Household listed as poor household
* Not involved with any government/non-government microfinance programme
* Not participants of any IYCF programme

Exclusion Criteria:

• Children with Severe Acute Malnutrition (SAM) or LAZ < -3SD of reference as per guideline

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 410 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Length for age Z-score (LAZ) | 12 months
  difference of 0.4 SD in LAZ between intervention and control group

SECONDARY OUTCOMES:
weight for age Z-score (WAZ) | 12 months
  Difference in mean weight for age Z-score (WAZ) of the children between intervention and control group at endline

CONTACTS AND LOCATIONS:
Overall Officials: Gulshan Ara, M.Sc, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Community, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ara G, Sanin KI, Khanam M, Sarker MSA, Tofail F, Nahar B, Chowdhury IA, Boitchi AB, Gibson S, Afsana K, Askari S, Ahmed T. A comprehensive intervention package improves the linear growth of children under 2-years-old in rural Bangladesh: a community-based cluster randomized controlled trial. Sci Rep. 2022 Dec 19;12(1):21962. doi: 10.1038/s41598-022-26269-w. PMID 36536016